CLINICAL TRIAL: NCT00002255
Title: An Open-Label Phase I/II Study of Recombinant Granulocyte Colony Stimulating Factor (r-metHuG-CSF) and Recombinant Erythropoietin (rHuEPO) Given Subcutaneously Along With Zidovudine (AZT) to Patients With the Acquired Immune Deficiency Syndrome (AIDS) or Severe AIDS-Related Complex (ARC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 077A; G-CSF 8808
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1991-01

CONDITIONS: HIV Infections
Keywords: Erythropoietin; Granulocyte Colony-Stimulating Factor; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Filgrastim; Epoetin Alfa; Zidovudine

INTERVENTIONS:
Drug: Filgrastim
Drug: Epoetin alfa
Drug: Zidovudine

SUMMARY:
To evaluate the safety, tolerance, and biological activity of filgrastim (recombinant granulocyte colony stimulating factor; G-CSF) given by daily subcutaneous injection prior to and concomitantly with erythropoietin (EPO) and zidovudine (AZT) in patients with AIDS or severe ARC. To evaluate the safety, tolerance, and biological activity of recombinant EPO given three times weekly by subcutaneous injection concomitantly with G-CSF and prior to and concomitantly with AZT in patients with AIDS or severe ARC. To study the safety and tolerance of three dose levels of AZT given concomitantly with G-CSF and EPO in patients with AIDS or severe ARC. To study the effects of G-CSF on neutrophil function and number in patients with AIDS or severe ARC. To study the effect of G-CSF alone and in combination with EPO on HIV replication in vivo as measured by circulating HIV p24 antigen, plasma HIV viremia, and semiquantitative HIV cocultures.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Ganciclovir (DHPG) for treatment of CMV infections.

Concurrent Treatment:

Allowed:

* Radiotherapy or laser therapy for Kaposi's sarcoma lesions provided dose does not exceed 3000 rads to any one lesion group and/or greater than 10 cm total body surface area.

Patients must have:

AIDS or severe ARC.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Opportunistic infection requiring ongoing therapy with known bone marrow-suppressive agents. (Exception:
* patients may take ganciclovir for treatment of CMV infections.)
* Evidence of a primary hematologic or infectious disorder unrelated to infection with the HIV virus.
* HIV-related dementia or altered mental status that would prohibit informed consent.
* More than 50 cutaneous Kaposi's sarcoma lesions or progression of Kaposi's sarcoma during the previous 30 days.
* Uncontrolled hypertension (defined as diastolic greater than 100 mm Hg).
* Presence of iron deficiency anemia as defined by serum ferritin less than 30 ng or iron TIBC ration less than 15 percent.

Concurrent Medication:

Excluded:

* Known bone marrow-suppressive agents such as trimethoprim / sulfamethoxazole or Fansidar for PCP prophylaxis.
* Any other non-FDA approved agent that may have antiretroviral activity.
* Hyperimmunization with polio virus, ribavirin, isoprinosine, dextran sulfate, fu zheng herbs, AL 721 or its congeners, imuthiol, interferons, chronic (> 10 days out of 30 days) use of Zovirax (acyclovir), and/or > 3 g/day oral vitamin C.

Patients with the following prior conditions are excluded:

* History of malignancy other than Kaposi's sarcoma.
* History of cardiovascular disease or seizures.

Prior Medication:

Excluded:

* Systemic cytotoxic chemotherapy within the previous 4 weeks for Kaposi's sarcoma.
* Investigational drugs within the previous 4 weeks.
* Prior colony stimulating factor (CSF).
* Any non-FDA approved drug within the previous 2 weeks.

Prior Treatment:

Excluded:

* Radiotherapy within the previous 4 weeks for Kaposi's sarcoma. Regular excessive use, currently or within the previous 3 months, of alcohol or hallucinogens or other psychotropic agents that are possibly addictive.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Miles SA, Study Chair; Slamon D, Study Chair
Locations (1):
- UCLA Med Ctr, Los Angeles, California, United States

REFERENCES:
- [Background] Miles SA, Mitsuyasu RT, Moreno J, Baldwin G, Alton NK, Souza L, Glaspy JA. Combined therapy with recombinant granulocyte colony-stimulating factor and erythropoietin decreases hematologic toxicity from zidovudine. Blood. 1991 May 15;77(10):2109-17. PMID 1709368